CLINICAL TRIAL: NCT02207881
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Topical VDO for the Treatment of Herpes Simplex Labialis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Collaborators: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YSP-RMN3001-01
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2014-07

CONDITIONS: Herpes Labialis
Keywords: herpes labialis; cold sore
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo gel, 25mg, 3 times up to 10 days
  Interventions: Drug: placebo
- VDO gel (Experimental): VDO gel 25mg, 3 times a day up to 10 days
  Interventions: Drug: VDO gel

INTERVENTIONS:
Drug: VDO gel — VDO gel
  Other Names: RMN3001
  Arms: VDO gel
Drug: placebo — matching placebo gel
  Other Names: RMN3001 placebo
  Arms: placebo

SUMMARY:
Recurrent herpes labialis are usually a minor malady of limited duration, although they are often painful and are uniformly discomforting for patients. Oral antivirals represent an advance in the treatment of recurrent herpes labialis, but the clinical implications are modest. Randomized, controlled clinical trials have shown that oral antivirals decrease the duration of lesion episodes and pain by approximately one day. In recurrent HSV infections including herpes labialis, many instances of viral re-activation occur without symptoms, and can only be identified by detection of virus on the lips of infected individuals. In these cases, the virus is cleared from the local site without the development of a classical ulcerative herpes lesion. In the other cases, the triggered specific immune response rapidly stops viral replication in the skin and also causes the development of the herpes lesion prodrome and a considerable part of the symptoms associated with a classical ulcerative herpes lesion. One could therefore predict that treatment with an antiviral drug alone would help the immune system in shortening the virus replication, but may not substantially reduce the disfiguring symptoms caused by the immune reaction. In dermatology, the principle of using an anti-inflammatory drug improve clinical outcomes by reducing inflammation-related symptoms associated with the infection has been well established. We have found that a topical formulation of VDO is useful for alleviating pain and inflammation associated with infection caused by herpes virus.

DETAILED DESCRIPTION:
In the treatment of oral herpes labialis, it is desirable to have local absorption of the drug to provide pain relief directly at the lesion sites while minimizing overall exposure.

The present study is designed to elucidate the effects of VDO ( on recurrent herpes simplex labialis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female in the age group 20 to 75 years old.
* History of recurrent herpes labialis with at least one recurrence occurred during the past twenty-four months.
* Onset of prodrome, erythema or vesicle within 72 hours of initiation of treatment with the study drug.
* Subjects with previous herpes simplex labialis episodes must be healed for at least 14 days before the baseline.
* Must be willing and able to participate and to provide written informed consent.
* Female subjects of childbearing potential must have a negative pregnancy test at screening and agree to use a proper contraceptive method during the study.

Exclusion Criteria:

* Women during pregnancy, lactation or breastfeeding.
* Subjects using topical steroids on or near the face or systemic (oral, intravenous) steroids within 7 days prior to study drug administration; use of inhaled or nasal spray steroids does not exclude a subject from the study.
* Subjects have used anti-viral agents or NSAID in the preceding 7 days.
* Subjects are unwilling to stop for using topical medical, OTC, cosmetic or facial skin care products in or around the oral area during the study period.
* Subjects with immunodeficiency disorders such as human immunodeficiency virus (HIV) infection or receiving cancer chemotherapy.
* Subjects who have a history of hypersensitivity to diclofenac, lidocaine or propylene glycol.
* Subjects who have a known hypersensitivity to local anesthetics of the amide type, diclofenac, aspirin, or other NSAIDs.
* Subjects who are taking antiarrhythmics drug during screening visit；
* Subjects who have a history of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs.
* Subjects who use during the perioperative period in the setting of coronary artery bypass graft (CABG) surgery within 6 months before the study drug using.
* Subjects have history of substance abuse or psychiatric illness that would preclude compliance with the protocol.
* Subjects who have serious, unstable, or clinically significant medical or psychological conditions, which, in the opinion of the investigator(s), would compromise the subject's participation in the study (including clinically significant dehydration or unstable vital signs).
* Subjects taking or having taken any other experimental drugs, drugs not approved in Taiwan, or participating in or having participated in other clinical studies in the 30 days prior to this clinical trial.
* Subjects who are considered unreliable as to medication compliance or adherence to scheduled appointments, or inappropriate for inclusion determined by the investigators.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adverse event | at the end of treatment (up to 10 days)
  Incidences of adverse event

SECONDARY OUTCOMES:
the duration and severity of pain | At the end of treatment (up to 10 days)
  Pain intensity will be measured at baseline and in the Subject's DRC on a daily basis while receiving study drug until end of study. Pain and itching assessments will be using a Visual Analogue Scale (VAS) ranging 0 (no pain/itching) to 10 (the worst pain/itching imaginable).
  The subject will be asked the following question exactly as follows：「On a scale 1 to 10 where 0 means on pain/itching, and 10 means the worst possible pain/itching, rate the worst pain/itching that you have since last assessment」

CONTACTS AND LOCATIONS:
Overall Officials: HUNG-MING WU, MD, PhD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan